CLINICAL TRIAL: NCT04905628
Title: Performance of the Dexcom Continuous Glucose Monitoring (CGM) System in Pregnant Women With Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-904284
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Dexcom CGM System: Dexcom CGM System
  Interventions: Device: Dexcom CGM System

INTERVENTIONS:
Device: Dexcom CGM System — Dexcom CGM System

SUMMARY:
Performance of the Dexcom Continuous Glucose Monitoring (CGM) System in Pregnant Women With Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed pregnancy
* Diagnosis of Gestational Diabetes (GDM), Type 1 Diabetes Mellitus (T1DM), or Type 2 Diabetes Mellitus (T2DM)
* Willing to wear up to the required number of Systems for the total duration of study wear
* Able to follow study procedures;
* Able to speak, read, and write in English or Spanish.

Exclusion Criteria:

* Extensive skin changes/diseases that preclude wearing the required number of Systems at the proposed wear sites
* Known allergy to medical-grade adhesives
* Hematocrit outside specification
* Prescribed drugs for treatment of pre-term labor or experiencing high-risk pregnancy complications during current pregnancy
* Currently receiving dialysis treatment or planning to receive dialysis during the sensor wear period
* Currently using Hydroxyurea for treatment
* Require a Magnetic Resonance Imaging (MRI) scan, Computed Tomography (CT) scan, or diathermy during the sensor wear period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 1. Age ≥ 18 years
  2. Confirmed pregnancy
  3. Diagnosis of Gestational Diabetes (GDM), Type 1 Diabetes Mellitus (T1DM), or Type 2 Diabetes Mellitus (T2DM)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Dexcom Continuous Glucose Monitoring (CGM) System Performance | 10 Days
  The Dexcom Continuous Glucose Monitoring (CGM) System performance will be assessed compared to Yellow Springs Instrument (YSI) comparator venous plasma measurements

SECONDARY OUTCOMES:
System Related Adverse Device Effects | 10 Days
  The Dexcom Continuous Glucose Monitoring (CGM) System will be characterized by Adverse Device Effects experienced by study participants

CONTACTS AND LOCATIONS:
Overall Officials: Carol Levy, MD, CDCES, Principal Investigator — Icahn School of Medicine at Mount Sinai; Sarit Polsky,, MD, MPH, Principal Investigator — Barbara Davis Center; Florence Brown, MD, Principal Investigator — Joslin Diabetes Center; Kristin Castorino, DO, Principal Investigator — Sansum Diabetes Research Institute; Amy Valent, DO, Principal Investigator — Oregon Health and Science University
Locations (5):
- United States (5):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Joslin Diabetes Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Polsky S, Valent AM, Isganaitis E, Castorino K, O'Malley G, Beck SE, Gao P, Laffel LM, Brown FM, Levy CJ. Performance of the Dexcom G7 Continuous Glucose Monitoring System in Pregnant Women with Diabetes. Diabetes Technol Ther. 2024 May;26(5):307-312. doi: 10.1089/dia.2023.0516. Epub 2024 Mar 1. PMID 38315503